CLINICAL TRIAL: NCT05437198
Title: Study of Microbiological Diversity in Exhaled Air in Adult Subjects With Chronic Obstructive Pulmonary Disease (COPD) and Subjects Free of COPD
Brief Title: Study of Microbiological Diversity in Exhaled Air in COPD and Free of COPD
Acronym: EXHALBIO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: EXHALBIO
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Obstructive Pulmonary Disease (COPD): Patients with chronic obstructive pulmonary disease will be recruited from the pulmonology or occupational pathology department. They are either active smokers or ex-smokers. They are over 18 years old
  Interventions: Other: collection of human exhalation
- NO-Chronic Obstructive Pulmonary Disease: The no-COPD are controls followed in chi créteil for another pathology. They are between 18 and 30 years old and 45 and 70 years old.
  They are either:
  * Ex-smoker
  * Active smoker
  * Non-smoker
  Interventions: Other: collection of human exhalation

INTERVENTIONS:
Other: collection of human exhalation — the collection of the exhalation will be carried out with a non-invasive device manufactured by a Chinese company.
  The collection of exhalation consists of the subject inhaling through the nose and exhaling gently through the mouth through a plastic straw for a time set at 5 min in the device

SUMMARY:
COPD and non-COPD patients will be included in the study after collection of their non-objection. The exhalation will be collected to study the microbiological diversity of human exhalations.

a second collection for the year +1 will be made, at the same time (between October and March).

DETAILED DESCRIPTION:
The subjects will be recruited during a medical visit in the Departments of Pneumology and Occupational and Environmental Pathologies.

After information and inclusion of the subject in the study, a collection of clinical data, the state of health and the smoking status of the subject will be carried out by the clinical study technician.

A collection of the exhalation will also be carried out by the clinical study technician.

Several groups of subjects will be formed according to pathologies (COPD versus non-COPD), age and smoking status

ELIGIBILITY:
Inclusion Criteria:

For COPD:

* Patients with chronic obstructive pulmonary disease
* Age: over 18

For non-COPD

* Absence of chronic obstructive pulmonary disease
* Age: between 18 and 30 years old and between 45 and 70 years old

Exclusion Criteria:

* Taking certain medications in the month preceding the sample (antibiotics, systemic corticosteroids, immunosuppressants)
* Person under guardianship or curatorship
* Pregnant or breastfeeding women
* Person unable to express his/her opposition, person deprived of liberty
* Existence of a chronic infectious pulmonary pathology such as (dilation of the bronchi, cystic fibrosis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with chronic obstructive pulmonary disease (COPD) and no-COPD control subjects
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number and dominant bacterial species in human exhalations of COPD subjects and non-COPD subjects | Baseline
  number and bacterial species

SECONDARY OUTCOMES:
Number and dominant bacterial species in human exhalations according to smoking status | Baseline
  number and bacterial species
Number and dominant bacterial species in human exhalations according to age | Baseline
  number and bacterial species
Number and dominant bacterial species in human exhalations for patients returning for consultation 1 year apart during the winter season | 1 year
  number and bacterial species

CONTACTS AND LOCATIONS:
Overall Officials: Jean Claude PAIRON, PhD, Principal Investigator — CHI créteil
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No